CLINICAL TRIAL: NCT04580953
Title: A Prospective Clinical Study Aimed to Assess the Technical Feasibility of RR2 Wearable Home Care Neuromodulation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv HealthCare Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CAR-POC-01
Record Dates: First submitted 2020-09-06; First posted 2020-10-09 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with CardiaCareTM RR2 (Experimental)
  Interventions: Device: CardiaCareTM RR2

INTERVENTIONS:
Device: CardiaCareTM RR2 — Treatment with CardiaCareTM RR2

SUMMARY:
RR2 is a medical, home-care, digital therapeutic, wearable device. Its main purpose is to deliver prescheduled, non-invasive, peripheral neuromodulation therapy, in conjunction with standard medical care, to relieve AF symptoms, recurrence and overall burden.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥18 with ECG documented and symptomatic recent onset atrial fibrillation (AF), lasting less than 48 hours
2. Symptoms related to AF with high probability
3. Recent conversion or cardioversion to normal sinus rhythm (NSR) as evident by a documented electrocardiograms (ECG)
4. Participants are able and willing to provide a signed informed consent
5. Participants are able and willing to use RR2 homecare device and wear an ECG patch or a Holter monitor for 24 hours.

Exclusion Criteria:

1. Hemodynamic instability (systolic blood pressure <100mmHg or heart rate >170 bmp)
2. An active myocardial infarction evident from ECG signs
3. Presence of pre-excitation syndrome
4. History of sick sinus syndrome
5. History of persistent AF with documented episodes of >7 days
6. Heart failure, acute or chronic
7. Participants currently enrolled in another study
8. Recurrent vaso-vagal syncopal episodes
9. Pregnancy or breast feeding
10. Pacemaker or Cardiac resynchronization therapy defibrillator (CRT-D) or any implantable electrical stimulating device
11. History of epilepsy or seizures
12. Peripheral neuropathy affecting the tested upper extremity
13. Participants unsuitable for participating in the study according to attending physician
14. Know allergy to .. (all materials that are in contact with patient's skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Assessment of system ECG function by the Number of ECG checks successfully conducted with record sent, received and stored by the system. | 8 weeks
  Number of ECG checks successfully conducted with record sent, received and stored by the system.
Assessment of system Nerumodulation function by the Number of self-treatments successfully conducted with record sent, received and stored by the system. | 8 weeks
  Number of self-treatments successfully conducted with record sent, received and stored by the system.

SECONDARY OUTCOMES:
Frequency of self-treatments during the treatment period | 8 weeks
  Number of self-treatments delivered by each patient throughout the 8-week period
Number of analyzed ECG | 8 weeks
  Number of analyzed ECG tests by cloud software
AF recurrence | 8 weeks
  Number of patients with symptomatic AF recurrence during the 8-week period
AFEQT quality of life questionnaire | 8 weeks
  Presence of AF-related symptoms and rate of significant symptom relief as assessed by AFEQT questionnaire
Centric questionnaire | 8 weeks
  Patient centric questionnaire
Unscheduled emergency department visits | 8 weeks
  Number of unscheduled emergency department visits due to atrial fibrillation
Number of patients with reduced premature atrial complexes (PAC's) and atrial runs | 8 weeks
  Number of patients with reduced premature atrial complexes (PAC's) and atrial runs from Week 1 to Week 8
Number of patients with acute reduction of PAC's 90 min | 8 weeks
  Number of patients with acute reduction of PAC's 90 min after each neuromodulation session
Heart rate variability (HRV) | 8 weeks
  Difference in acute heart rate variability (HRV) parameters before and after treatments
First AF event | 8 weeks
  Time from Baseline until first AF event
AF burden | 8 weeks
  AF burden measured as number of registered AF episodes
AF burden | 8 weeks
  AF burden measured as the longest AF episode

CONTACTS AND LOCATIONS:
Overall Officials: Avi Sabbag, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel